CLINICAL TRIAL: NCT05497635
Title: A Randomized,Double-blind, Placebo-controlled, Multiple Ascending-Dose Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of STSA-1002 Injection in Healthy Subjects
Brief Title: A Study of STSA-1002 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1002-03
Record Dates: First submitted 2022-08-01; First posted 2022-08-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Subject

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A low dose of group (Experimental): All subjects will be randomized to receive low dose of STSA-1002 or dose-matched placebo.
  Interventions: Drug: STSA-1002 Injection; Drug: Placebo
- A middle dose of group (Experimental): All subjects will be randomized to receive middle dose of STSA-1002 or dose-matched placebo.
  Interventions: Drug: STSA-1002 Injection; Drug: Placebo
- A high dose of group (Experimental): All subjects will be randomized to receive high dose of STSA-1002 or dose-matched placebo.
  Interventions: Drug: STSA-1002 Injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1002 Injection — Intravenous injection
Drug: Placebo — Intravenous injection

SUMMARY:
This study is a Phase Ib, randomized, double-blind, placebo-controlled, multiple dose, dose escalation safety, tolerability,pharmacokinetic and pharmacodynamic study of STSA-1002 injection in healthy subjects. A total of 26 healthy subjects were enrolled in three dosage groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, aged ≥ 18 but ≤ 45, male and female.
* Weight:Male≥50.0kg,Female≥45kg;Body mass index: 19.0-26.0 kg/m2, inclusive.
* Medical history, vital signs, physical examination, laboratory examination (including blood routine, urine routine, blood biochemistry, coagulation function test, etc.) and all tests related to the test were normal or abnormal as determined by the researcher and had no clinical significance.
* Subjects (including their partners) must take effective contraceptive measures and have no birth plan or sperm or egg donation plan during the trial period and within 6 months after the end of the last administration.
* Subjects are aware of the content, process and possible adverse reactions of the study and voluntarily signed the informed consent form(ICF).

Exclusion Criteria:

* History of tuberculosis; or combined with mixed lymphocyte culture + interferon assay results, chest imaging comprehensive evaluation of tuberculosis infection (if necessary, tuberculosis experts should be jointly evaluated).
* Any clinically serious diseases such as respiratory, circulatory, digestive, urinary, blood, endocrine, neurological or mental disorder, or a history of the above diseases or any other diseases or physiological conditions that can interfere with the test results.
* With any major surgical or surgical that possibly affects drug absorption, distribution, metabolism or excretion(Except appendicitis) within 2 months before screening or plan to undergo surgery during the study period.
* Subjects with allergies or allergies to any components of the investigational drug and its excipients(such as allergies to two or more drugs, food, pollen), or the IgE is higher than the upper limit of normal.
* Positive screening test results for human immunodeficiency virus (HIV) antibodies, syphilis-specific antibody, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCVAb).
* Subjects with abnormal blood white blood cell count and absolute neutrophil count during the screening period with clinical significance; or hemoglobin: male <120g/L or female <110g/L.
* Drug abuse within 1 year before screening [such as morphine, ketamine (K powder), THC (marijuana), methamphetamine (ice), MDMA (ecstasy) ), cocaine, etc.]; or positive urine screening for drug abuse.
* Subjects who have taken drugs that may affect immune function within 6 months before screening, have received any monoclonal antibody or biological agent for treatment (for any illness) within the previous 3 months, and have taken prescription drugs,non-prescription drugs,chinese herbal medicine within 14 days before screening.
* Alcoholism within 6 months before screening (drinking more than 14 units of alcohol per week: 1 unit = 285mL of beer, or 25mL of spirits, or 100mL of wine) or unable to stop consuming any alcoholic products after enrollment until the entire study period or a positive alcohol breath test result.
* Subjects who smoking (more than 5 cigarettes per day on average) within 3 months before screening or who could not stop using any tobacco products until the whole study period after enrollment.
* Subjects who drink too much (more than 8 cups a day, 1 cup = 200 mL) of tea, coffee and other beverages rich in xanthine within 3 months before screening, or food or beverages that affect drug absorption, distribution, metabolism, and excretion.
* Donation of blood or lost more than 400ml within 3 months before the first investigational product administration or plan to donate blood or blood components during the study period or within 3 months after the end of the study, or have a history of blood transfusion within 4 weeks before the first drug use of the study.
* Subjects who participated in any unmarked drug, vaccine or medical device clinical trial within 3 months before screening and applied the drug, vaccine or medical device in the trial.
* Vaccination within 14 days before the first dose or ready to be vaccinated during the study period to 2 months after the end of the study.
* Subjects who have used long-acting estrogen or progestogen injections or implants within 6 months before the study or those who have used short-acting contraceptives within 4 weeks before the study.
* Female subjects who have had unprotected sex within 14 days prior to screening.
* Blood β-HCG test positive or above the upper limit of the normal range (Female subjects).
* Pregnant or lactating.
* Any food or drink rich in xanthine (such as coffee, strong tea, chocolate, etc.) or food or drink that affects drug absorption, distribution, metabolism, and excretion within 48 hours before administration.
* Unable to follow a unified diet (such as special requirements for diet, intolerance to standard meals, etc.).
* Intolerance to venipuncturing blood collection, transfusion, or a history of blood and needle sickness.
* Other circumstances in which the researcher considers it inappropriate to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events、Clinically Significant Laboratory Abnormalities、Clinically Significant Electrocardiogram、Vital Signs And Physical Examination Abnormalities. | Up to Study Day 56
  To evaluate the safety and tolerability of multiple intravenous administration of STSA-1002 in healthy adult subjects.
Maximum plasma concentration (Cmax) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Area under the plasma concentration-time curve from time 0 to the collection time point t of the last measurable concentration (AUC0-t) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Time of maximum concentration (Tmax) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Elimination half-life (t1/2) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Mean residence time (MRT) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Clearance (CL) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Apparent volume of distribution (Vz) | From Day 0 to Day 56
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1002 in healthy adult subjects
Maximum Concentration of the Analyte in Plasma at steady state(Cmax, ss) | From Day 0 to Day 56
  To evaluate the multidose PK characteristics of STSA-1002 in healthy adult subjects
Minimum Measured Concentration of the Analyte in Plasma at Steady State(Cmin, ss) | From Day 0 to Day 56
  To evaluate the multidose PK characteristics of STSA-1002 in healthy adult subjects
Time-averaged concentration at steady state(Cav, ss) | From Day 0 to Day 56
  To evaluate the multidose PK characteristics of STSA-1002 in healthy adult subjects
Area under the concentration curve from time 0 extrapolate to infinite time(AUCinf,ss) | From Day 0 to Day 56
  To evaluate the multidose PK characteristics of STSA-1002 in healthy adult subjects
Degree of fluctuation(DF) | From Day 0 to Day 56
  To evaluate the multidose PK characteristics of STSA-1002 in healthy adult subjects
Accumulation factor | From Day 0 to Day 56
  To evaluate the multidose PK characteristics of STSA-1002 in healthy adult subjects

SECONDARY OUTCOMES:
Change from baseline in concentration of free C5a and anti-drug antibody | From Day 0 to Day 56
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1002 in healthy subjects
Change from baseline in concentration of Myeloperoxidase（MPO）、Neutrophil elastase（NE）、Proteinase3（PR3）、 C-X-C chemokine receptor 1(CXCR1) | From Day 0 to Day 56
  To evaluate the effect of STSA-1002 on MPO、NE、PR3、CXCR1

CONTACTS AND LOCATIONS:
Overall Officials: Xinghe Wang, Ph.D, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (2):
- China (2):
  - Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Of Xingtai Medical College, Xingtai, Hebei

IPD SHARING:
Plan to Share IPD: No